CLINICAL TRIAL: NCT04568902
Title: A Phase 1 Study of H3B-6545 in Japanese Women With Estrogen Receptor-positive, HER2 Negative Breast Cancer
Brief Title: Study of H3B-6545 in Japanese Women With Estrogen Receptor (ER)-Positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H3B-6545-J081-103
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasms
Keywords: H3B-6545; ER-positive; HER2-negative
MeSH Terms: conditions — Breast Neoplasms | interventions — H3B-6545; Histamine Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Part: H3B-6545 300 mg (Experimental): Participants will receive H3B-6545 300 milligram (mg) tablets, orally, once daily in 28 days cycle until disease progression, violation of study requirements, unable to continue study based on investigator opinion or withdrawal of consent.
  Interventions: Drug: H3B-6545
- Dose Escalation Part: H3B-6545 450 mg (Experimental): Participants will receive H3B-6545 450 mg tablets, orally, once daily in 28 days cycle until disease progression, violation of study requirements, unable to continue study based on investigator opinion or withdrawal of consent.
  Interventions: Drug: H3B-6545
- Antihistamine Prophylactic Administration Part (Experimental): Participants will receive prophylactic treatment with non-sedating systemic antihistamine, orally, once from Cycle 1 Day 1 until Cycle 1 Day 28, followed by H3B-6545 450 mg tablets, orally, once daily in 28 days cycle until disease progression, violation of study requirements, unable to continue study based on investigator opinion or withdrawal of consent.
  Interventions: Drug: H3B-6545; Drug: Antihistamine
- Randomization Part (Experimental): Participants will be randomized in 1:1 ratio to receive H3B-6545 450 mg, tablets, orally, once daily in 28 days cycle either with non-sedating systemic antihistamine prophylactic administration from Day 1 until Day 28 of Cycle 1 OR without antihistamine prophylactic administration until disease progression, violation of study requirements, unable to continue study based on investigator opinion or withdrawal of consent.
  Interventions: Drug: H3B-6545; Drug: Antihistamine

INTERVENTIONS:
Drug: H3B-6545 — H3B-6545 oral tablets.
Drug: Antihistamine — Systemic antihistamine oral drug such as fexofenadine, loratadine and cetirizine.
  Arms: Antihistamine Prophylactic Administration Part; Randomization Part

SUMMARY:
The purpose of study is to determine tolerability and safety profile of H3B-6545 in Japanese women with ER-positive, HER2-negative breast cancer, and also to confirm the dose applicability to Japanese.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a histologically and/or cytologically confirmed diagnosis of ER-positive, HER2-negative breast cancer.

   Note: Status of ER and HER2 should be diagnosed by method approved by regulatory authority
2. Only females, age greater than or equal to (>=) 20 years at the time of informed consent.
3. Prior therapy for breast cancer in the adjuvant and/or advanced/metastatic setting must have included a minimum of:

   1. two prior hormonal therapies, or
   2. one prior hormonal therapy and one prior chemotherapy regimen, or
   3. one prior hormonal therapy and a cyclin-dependent kinase (CDK4/6) inhibitor.
4. Participant has an ECOG-PS of 0 or 1.
5. Participant has adequate bone marrow and organ function, as defined by the following laboratory values:

   * Absolute neutrophil count (ANC) >=1.5*10˄9/liter (L).
   * Platelets >=100*10˄9/L.
   * Hemoglobin >=9.0 gram per deciliter (g/dL).
   * Potassium, sodium, calcium (corrected for serum albumin) and magnesium less than or equal to (<=) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
   * International normalized ratio (INR) <=1.5.
   * Serum creatinine <=1.5*upper limit of normal (ULN).
   * Serum albumin >=3.0 g/dL (>=30 gram per liter [g/L]).
   * Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) <=3.0*ULN. If the participant has liver metastases, ALT and AST <=5.0*ULN.
   * Total serum bilirubin less than (<) 1.5*ULN.
6. Participants who are expected to survive for 3 months or longer after starting administration of the investigational drug.
7. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Participant with inflammatory breast cancer.
2. Participant is currently receiving or has received systemic corticosteroids <=2 weeks prior to starting study drug, or has not fully recovered from side effects of such treatment.

   Note: The following uses of corticosteroids are permitted: inhaled sprays (example- for obstructive airways diseases), eye drops or local injections (example- intra-articular).
3. Washout period required from the end of prior treatment to the first administration of study drug will be as follows.

   1. Anti-cancer therapy

      * Antibody and other study drugs: greater than (>) 4 weeks (however, in the case where the half-life of other study drugs is known and 5*half-lives of that study drug is less than or equal to 4 weeks, participants can be eligible after >=5*half-lives of that study drug has passed).
      * Prior chemotherapy (except small-molecule targeted therapy), surgical therapy, radiation therapy: >3 weeks.
      * Endocrine therapy, immunotherapy (except antibody drug), small-molecule targeted therapy: >2 weeks.
   2. Supportive therapy • Blood/platelet transfusion, hematopoietic stimulating agent including granulocyte colony-stimulating factor (G-CSF) formulation: >2 weeks.
4. Participant has active cardiac disease or a history of cardiac dysfunction, including any of the following:

   1. History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry.
   2. History of documented congestive heart failure (New York Heart Association [NYHA] functional classification II to IV).
   3. Documented cardiomyopathy.
   4. Participant has a left ventricular ejection fraction (LVEF) <50 percent (%) as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO).
   5. History of any cardiac arrhythmias, example- ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
   6. Heart Rate <60 beats per minute (bpm) on the screening.
   7. On screening, any of the following cardiac parameters: PR interval >220 millisecond (msec), QRS interval >10˄9 msec, or QT interval with Fridericia's correction (QTcF) >450 msec.
   8. Systolic blood pressure (BP) not deemed clinically controlled by the investigator.
5. Participant has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of H3B-6545.
6. Participant has a known hypersensitivity to any of the excipients of H3B-6545.
7. Known to be human immunodeficiency virus (HIV) positive.
8. Active viral hepatitis (B or C) as demonstrated by positive serology. Participants with chronic hepatitis B virus (HBV) infection is on antiviral therapy is eligible.
9. Participant has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate participant participation in the clinical study (example- chronic pancreatitis, thyroid dysfunction etc).
10. Any adverse event related to previous therapies for breast cancer that has not resolved to <=Grade 1 (with exception of the alopecia).
11. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG] test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
12. Women of childbearing potential who don't agree that both the participant and her partner will use a medically effective method for contraception (as below) throughout the entire study period or for 28 days after study drug discontinuation.

    Note: Condom*, contraceptive sponge**, foam**, jelly**, diaphragm**, intrauterine device (IUD) *, or use of oral contraception* from at least 4 weeks before starting the study treatment (*Approved drugs or certified medical devices in Japan, **Non-approved drugs or certified medical devices in Japan) If a participant is on oral contraceptives, they should also be using some additional method.
13. Alcohol dependency within 6 months before study entry.
14. Participant has a concurrent malignancy or malignancy within 3 years of enrollment, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer.
15. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
16. Diagnosed with meningeal carcinomatosis.
17. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example- radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
18. Participant has a known intolerability to any oral antihistamine drug (only for Antihistamine Prophylactic Administration Part and Randomization Part).
19. Participant needs to receive systemic or topical usage of either antihistamine or corticosteroid during Cycle 1 (only for Randomization Part).

    Note: The following uses of corticosteroids are permitted: inhaled sprays (example, for obstructive airways diseases), eye drops or local injections (example, intra-articular).
20. Participants initiated to receive drugs may cause rash 7 days prior to starting study drug.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) | Up to Cycle 1 (each cycle length is equal to [=] 28 days)
  Toxicity will be assessed according to National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE), v5.0. DLT is defined as any of the following events occurred within the Cycle 1 of the administration of H3B-6545: Febrile neutropenia, Grade 4 neutropenia that does not resolve to Grade<=2 within 7days, Grade 4 thrombocytopenia, Grade3 thrombocytopenia>=7days or requiring platelet transfusion, Grade3 thrombocytopenia associated with bleeding, Grade4 anemia or Grade3 anemia requiring erythrocyte transfusion; Grade3 or 4 bilirubin increase, AST or ALT>=10*ULN which does not resolve to Grade2 or less within 7days and/or else is clinically significant; Non-hematological toxicities Grade4 and Grade3 with exception of abnormal clinical laboratory values with no clinical significance and events which can be managed and controlled to Grade2 or less by maximal medical management within 7days, participant administered<70% of prescribed dose due to intolerable toxicity.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to 36 months
Percentage of Participants With Incidence of Rash | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in Laboratory Values | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in Vital Sign Values | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in Weight Values | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in Physical Examinations | Baseline up to 36 months
Number of Participants With Clinically Significant Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG-PS) | Baseline up to 36 months
  ECOG performance score is measured on 6 point scale to assess participant's performance status, where: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; Grade 5: Dead.

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
Tmax: Time of Maximum Observed Plasma Concentration of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
AUC 0-t: Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
Rac: Accumulation Ratio of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
AUC 0-inf: Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
T1/2: Terminal Half-life of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
CL/F: Apparent Total Body Clearance of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)
Vz/F: Apparent Volume of Distribution at Terminal Phase of H3B-6545 | Dose Escalation and Antihistamine Prophylactic Administration Part: Cycle 1 Days 1 and 15: 0-24 hours post dose; Randomization Part: Cycle 1 Days 1 and 15: 0-6 hours post dose (cycle length=28 days)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Eisai Trial Site 2, Chūōku
  - Eisai Trial Site 1, Kōtoku

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Furman C, Puyang X, Zhang Z, Wu ZJ, Banka D, Aithal KB, Albacker LA, Hao MH, Irwin S, Kim A, Montesion M, Moriarty AD, Murugesan K, Nguyen TV, Rimkunas V, Sahmoud T, Wick MJ, Yao S, Zhang X, Zeng H, Vaillancourt FH, Bolduc DM, Larsen N, Zheng GZ, Prajapati S, Zhu P, Korpal M. Covalent ERalpha Antagonist H3B-6545 Demonstrates Encouraging Preclinical Activity in Therapy-Resistant Breast Cancer. Mol Cancer Ther. 2022 Jun 1;21(6):890-902. doi: 10.1158/1535-7163.MCT-21-0378. PMID 35642432